CLINICAL TRIAL: NCT03516916
Title: Surviving Rectal Cancer at the Cost of a Colostomy International Validation of the Colostomy Impact Score
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Aarhus University Hospital (Other)
Collaborators: Eloy Espin, Department of Surgery, Universidad Autonoma de Barcelona (Unknown); Kelly Buzatti, Federal University of Minas Gerais (Unknown); Dong Pang, Peking University School of Nursing (Unknown); Mansoura University (Other); Edgar Furnee, University Medical Center, Groningen (Unknown); Annika Sjövall, Karolinska Institute, Stockholm (Unknown); Tomas Poskus, Faculty of Medicine, Vilnius University (Unknown); Sheba Medical Center (Other Government); Andrea Warwick, Redcliffe and QEII Jubilee Hospitals (Unknown); Nuno Rama,Centro Hospitalar Leiria Pombal (Unknown)
Responsible Party: Principal Investigator, Helle Ø Kristensen, MD, Aarhus University Hospital
Other Study IDs: 490-98-0860
Record Dates: First submitted 2018-04-24; First posted 2018-05-07 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Rectal Neoplasms; Quality of Life; Colostomy Stoma
Keywords: Rectal cancer, HRQoL, Stoma, Colostomy, Patient reported outcome measure (PROM)
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (15):
- Australia: Patients with a permanent colostomy after curative surgery for rectal cancer
  Interventions: Other: Questionnaires on HRQoL and sociodemography
- Brazil: Patients with a permanent colostomy after curative surgery for rectal cancer
  Interventions: Other: Questionnaires on HRQoL and sociodemography
- China: Patients with a permanent colostomy after curative surgery for rectal cancer
  Interventions: Other: Questionnaires on HRQoL and sociodemography
- Denmark: Patients with a permanent colostomy after curative surgery for rectal cancer
  Interventions: Other: Questionnaires on HRQoL and sociodemography
- Egypt: Patients with a permanent colostomy after curative surgery for rectal cancer
  Interventions: Other: Questionnaires on HRQoL and sociodemography
- Israel: Patients with a permanent colostomy after curative surgery for rectal cancer
  Interventions: Other: Questionnaires on HRQoL and sociodemography
- Lithuania: Patients with a permanent colostomy after curative surgery for rectal cancer
  Interventions: Other: Questionnaires on HRQoL and sociodemography
- the Netherlands: Patients with a permanent colostomy after curative surgery for rectal cancer
  Interventions: Other: Questionnaires on HRQoL and sociodemography
- Portugal: Patients with a permanent colostomy after curative surgery for rectal cancer
  Interventions: Other: Questionnaires on HRQoL and sociodemography
- Russia: Patients with a permanent colostomy after curative surgery for rectal cancer
  Interventions: Other: Questionnaires on HRQoL and sociodemography
- South Africa: Patients with a permanent colostomy after curative surgery for rectal cancer
  Interventions: Other: Questionnaires on HRQoL and sociodemography
- Spain: Patients with a permanent colostomy after curative surgery for rectal cancer
  Interventions: Other: Questionnaires on HRQoL and sociodemography
- Sweden: Patients with a permanent colostomy after curative surgery for rectal cancer
  Interventions: Other: Questionnaires on HRQoL and sociodemography
- Turkey: Patients with a permanent colostomy after curative surgery for rectal cancer
  Interventions: Other: Questionnaires on HRQoL and sociodemography
- the United Kingdom: Patients with a permanent colostomy after curative surgery for rectal cancer
  Interventions: Other: Questionnaires on HRQoL and sociodemography

INTERVENTIONS:
Other: Questionnaires on HRQoL and sociodemography — All patients are asked to answer a panel of questionnaires to test validity and reliability of the Colostomy Impact Score.

SUMMARY:
The formation of a colostomy following surgery for rectal cancer changes body image, challenges patient practical skills and threatens quality of life. As the oncological results have improved over the last decades the number of survivors from rectal cancer who have to adjust to a cancer free life in their own homes is increasing. To enable the identification of the patients with stoma-related reduced health-related Quality of life (HRQoL) in a quick and reliable way we recently developed the Colostomy Impact Score (CI-score) comprising 7 items of stoma related factors with significant impact on HRQoL. The purpose of the present project is to perform an international validation of the CI-score and to demonstrate its applicability.

The construct validity of the CI-score will be studied internationally on crosssectional cohorts of patients with permanent colostomy after abdominoperineal excision (APE) or Hartmann's procedure in Denmark, Sweden, Spain, the Netherlands, United Kingdom, Turkey, Brazil, Egypt, Russia, Lithuania, Israel, Portugal, South Africa, Australia and China. This will be done by testing the CI-score against five anchor questions stoma impact on HRQoL, the 5 Level version og the EuroQol measuer (EQ-5D-5L) and version 3.0 of the Quality of Life Questionnaire from the European Organisation for Research and Treatment of Cancer (EORTC QLQ C30 questionnaire v3.0).

The impact of the challenges related to having a stoma may vary with different demographic, socioeconomic and cultural factors. Supplementary data on stoma care, demographics and socioeconomic status will be gathered to study the impact of patient-related factors and cultural differences on HRQoL in rectal cancer survivors with an ostomy.

DETAILED DESCRIPTION:
This retrospective cohort study has three main aims: 1) To identify demographic and socioeconomic factors influencing stoma impact and HRQoL, 2) To asses reliability and to validate the translated and cross-cultural adapted CI score internationally in multiple different centres, across a variety of patient groups and across cultural, religious, socioeconomic and physical borders and 3) To investigate if differences in everyday stoma care and -costs across countries and cultures affect CI or HRQoL.

International validation will be conducted as a retrospective cohort study on patients with a permanent colostomy after curative intended surgery more than 12 months prior to inclusion. Local health care professionals will identify includable patients and register relevant clinical information on each patient from the hospital chart. Most centres will include patients from national or regional databases, some will however include conveniently if a database is not available. Our international collaborators will be responsible for sending out and collecting the questionnaires and returning the completed questionnaires to the undersigned. In countries with sufficient internet accessibility and -infrastructure the data collection will be web based i.e. patients are sent a link to the redcap-database for them to enter their answers directly. Some centres will employ paper versions of the questionnaires. In areas with substantial number of illiterates investigator led interviews can be performed.

As the CI-score is a construct based on a formative model, statistical analysis based on the Classical Test Theory(CCT) and Item Response Theory (IRT) cannot be applied. However, the following aspects of validity and reliability from the Consensus-based Standards for the selection of health Measurement Instruments (COSMIN) checklist15-17 can and will be evaluated:

Content validity: Comprehensiveness and relevance of the questions in the CI-score have been ensured with the way of the development of the CI-score with the starting point in a Basic Stoma Questionnaire developed by an expert group supplemented by patients ensuring that all possible factors affecting stoma function/impact was included before regression analysis lead to the seven weighed questions1. After translation and cross-cultural adaptation face-validity of each translated CI-score will be assessed again by the collaborators before inclusion of patients.

Construct validity: This will be tested with hypothesis-testing. Hypotheses regarding mean differences and expected correlations between scores of instruments are formulated a priori. Hypotheses on how the CI-score and HRQoL are related to other factors are formulated a priori. For convergent validation the CI-score will be tested against 5 anchor questions (not validated) and the EORTC QLQ C30+ the colorectal specific CR29 (validated). Cross-cultural validity: See translation section.

Reliability: For a randomly selected subgroup in each country the CI-score and anchor question will be administered twice with an interval of approximately 2 weeks. The two administrations will be independent and both the setting when answering and the forms of administration will be similar for the individual patient. For ensuring stable patients an extra question on recent changes in stoma function will be added to the retest.

Translation of the CI-score will be managed by the lead institution with few exceptions (Turkey, Russia, Israel) and will follow the translation procedure recommended by the World Health Organization. All translations are produced by a forward-backward procedure. The latter procedure is performed to ensure, that the original meaning of the concepts is derived.

The original Danish version of the CI-score has already undergone a professional translation to English. A professional translation agency will perform the translation of the English version to languages in the included countries. All questionnaires/Case Report Forms (CRF) to be filled in by patients will undergo the same translation procedure as above.

A master version of the questionnaires will be collected into a booklet. On this basis, a RedCap database will be constructed to allow for direct electronic data entry by patients. Patient not able to access the web-based system, will fill in a paper version of the booklet. According to variation between populations in respect to practically illiterate's investigator lead data collection will be allowed. However, this should be agreed by the local investigation and the steering group in the planning of the data collection and included as individual amendment to the final protocol.

Data analysis:

Construct validity: Convergent validity will be studied by testing the CI-score on APE/Hartmann-patients against two measures of HRQoL; the anchor-questions assessing the overall stoma-impact on HRQoL, the EORTC QLQ C30 questionnaire version 3.0 and the EORTC QLQ CR29. Construct validity will furthermore be assessed by hypothesis-testing assessing the direction and magnitude of the expected correlations. Test-retest reliability will be studied on a subgroup in all included countries. Also, we will include questions on background demographics, socioeconomic status, everyday stoma care and -costs thereby enabling investigation of the practical and economic aspect of living with a stoma varying from country to country.

Statistical analysis:

Statistical analysis will be performed separately for each country. The correlations between total CI-score, anchor questions and the EORTC questionnaire results will be calculated for all participating patients according to the guidelines for the scores. For each CI-score group (minor CI/major CI) the mean EORTC QLQ C30-score will be calculated, testing the overall difference of impact on HRQoL between the CI-score groups.

Using the anchor-questions, the patients are divided into two HRQoL groups of those reporting no/minor or some/major impact on HRQoL. Relationship between CI-score and HRQoL group will be illustrated in box-plot for each country, where we expect statistically significant differences in median CI-score between the two HRQoL groups. Differences will be tested by Mann-Whitney U test. A contingency 2 by 2 table will be used to assess the degree of agreement between the two CI-score groups and the two HRQoL groups. Based on this, the sensitivity for the score will be calculated for each country. The added questions about irrigation and stoma-bag change frequency will be compared country-wise. Univariate regression analysis, descriptive analysis and estimation of impact on HRQoL will be performed. Test-retest reliability will be evaluated using Intraclass Correlation Coefficient and Cohens' Kappa.

ELIGIBILITY:
Inclusion Criteria:

* Curative intended Hartmann's procedure or abdominal perineal excision >12 months ago for carcinoma of the rectum
* Permanent colostomy

Exclusion Criteria:

* Age < 18 years
* Recurrence of cancer
* Mental dementia
* Unable to understand the actual language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a permanent colostomy after curative intended surgery for rectal cancer. Time since surgery must be more than 1 year. In some countries the cohort will be extracted from a national or institutional registry representing all operated patients in a certain time period that allows for inclusion of 250 patients. In countries whithout such registries convenient inclusion from the surgical department or stoma clinic.
Sampling Method: Non-Probability Sample
Enrollment: 3750 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Validity of the Colostomy Impact Score | The end of 2018
  Description of sensitivity, specificity and construct validity (hypothesis testing) of the Colostomy Impact Score.
Impact of demographic, socioeconomic and religious factors on HRQoL in rectal cancer survivors with a colostomy | The end of 2018
  Comparing HRQoL between sexes, age groups and different socioeconomic and religious groups and by country.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Ø Kristensen, MD, Principal Investigator — Danish Cancer Society Centre for Research on Survivorship and Late Adverse Effects After Cancer in the Pelvic Organs, Department of Surgery, Aarhus University Hospital
Locations (1):
- Department of Surgery, Aarhus University Hospital, Aarhus, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT03516916/Prot_SAP_001.pdf